CLINICAL TRIAL: NCT04537091
Title: Radial Extracorporeal Shock Wave Therapy Versus Platelet-rich Plasma Injection for the Treatment of Greater Trochanteric Pain Syndrome With Gluteal Tendinopathy: a Randomized Controlled Trial
Brief Title: Radial Extracorporeal Shock Wave Therapy Versus Platelet-rich Plasma Injection for Greater Trochanteric Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Mustafa Corum, Principal Investigator, Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2020-309
Record Dates: First submitted 2020-08-21; First posted 2020-09-03 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2020-09

CONDITIONS: Gluteal Tendinopathy; Greater Trochanteric Pain Syndrome

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESWT group: rESWT (Experimental): rESWT treatment was applied to patients
  Interventions: Procedure: rESWT
- PRP group: PRP injection (Experimental): PRP treatment was applied to patients
  Interventions: Procedure: PRP injection

INTERVENTIONS:
Procedure: rESWT — rESWT was administered once per week for 3 weeks with 4 bar pneumatic pressure, 10 Hz frequency, with 2000 pulses. Radial shock waves were transmitted to the greater trochanteric region with the maximum pain/tenderness that was identified with patients' reaction with small circular movements with an adequate amount of contact gel
  Arms: ESWT group: rESWT
Procedure: PRP injection — PRP injection is performed with a high resolution 7-12-megahertz linear probe ultrasonography device. 15 ml of blood will be drawn from the patients and the blood will be centrifuged for 5 minutes. 4-5 ml PRP will be injected into the affected gluteal tendons accompanied by ultrasonography.
  Arms: PRP group: PRP injection

SUMMARY:
Greater trochanteric pain syndrome (GTPS), is characterised by pain around the greater trochanter. Failure of first-line management for GTPS is followed by second-line treatments range from extracorporeal shock wave therapy (ESWT), corticosteroid or platelet-rich plasma (PRP) injections, and surgery. In a systematic reviews, PRP seems a viable effective and safe alternative option for GTPS after failed physical therapy. Also, positive results from previous systematic reviews involving radial ESWT (rESWT) as a treatment for GTPS.

In the literature review, there is no comparison of the effectiveness of ESWT and PRP injection in patients with GTPS. The aim of this study was to investigate the effects of rESWT and PRP injection on pain, hip disability, and quality of life in patients with GTPS

DETAILED DESCRIPTION:
The pain and activities of daily living, referring to the previous week, and assessments of hip function (limping) and range of motion were evaluted by Harris Hip Score (HHS). The pain severity during rest and activity in the previous week was evaluted by Visual Analog Scale (VAS). The pain and activity limitation was evaluted by The Roles and maudsley (RM). The quality of life was evaluted by The EQ-5D-3L scale.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* Complaining of pain located anterior, lateral or posterior to the great trochanter for more than 3 months
* Pain while lying on the affected side
* Local tenderness on palpation of the area of the great trochanter
* MRI evidence of gluteus minimus or medius tendinopathy
* Refractory to conservative management

Exclusion Criteria:

* Presence of signs and symptoms of another cause of regional hip pain.
* Full-thickness tear of the involved gluteal tendons, bursa, and intra-articular structures
* Evidence of concomitant injury to the involved lower extremity, including radiculopathy or radiculitis, ischial tuberosity avulsion
* Severe knee or hip osteoarthritis
* Previous hip surgery or use of ESWT for GTPS.
* Acute low back pain
* Implanted pacemaker
* Vascular, neurologic, rheumatic diseases.
* Any neoplastic disorders
* Blood coagulation disorders or use of antiplatelet or anticoagulant drugs
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-01-05 (Actual)

PRIMARY OUTCOMES:
Harris Hip Score (HHS) | Changes from baseline in Harris Hip Score to 1 month and 6 months.
  The index consists of questions about pain and activities of daily living, referring to the previous week, and assessments of hip function (limping) and range of motion. Score ranges from 100 (no disability) to 0 (maximum disability).

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) | Changes from baseline in Visual Analog Scale score to 1 month and 6 months.
  The self-evaluation of pain severity during rest and activity in the previous week was calculated using a 10-cm VAS scale, where 0 in the left corner of the scale represented 'no pain' and 10 in the right corner represented 'the worst pain that could be imagined'
The Roles and maudsley (RM) | Changes from baseline in Roles and maudsley score to 1 month and 6 months.
  RM score was used to evaluate pain and activity limitation as classified in four categories: 1 point = excellent, 2 points = good, 3 points = fair, and 4 points = poor.
EuroQol five-dimensional questionnaire (EQ-5D-3L) | Changes from baseline in EuroQol five-dimensional questionnaire score to 1 month and 6 months.
  The EQ-5D-3L scale, which scores five health conditions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) through evaluation at 3 levels (no problems, some problems, or extreme problems), was used to evaluate the quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Corum, MD, Study Chair — Istanbul Physical Medicine Rehabilitation Training & Research Hospital
Locations (1):
- Istanbul Physical Medicine and Rehabilitation Training and Research Hospital, Istanbul, Bahcelievler, Turkey (Türkiye)